CLINICAL TRIAL: NCT02441296
Title: Postprandial Serum Responses to Various Infant Formulas and Breast Milk in Infants- a Pilot Study
Brief Title: Carbohydrate and Metabolism: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: University of California, Davis (Other); Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2013-152-31M
Record Dates: First submitted 2015-04-08; First posted 2015-05-12 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Infant; Metabolism
MeSH Terms: interventions — Food, Formulated; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Formula with lactose (Experimental): Carbohydrate-free formula with added lactose
  Interventions: Other: Formula with lactose
- Formula with maltodextrins (Experimental): Carbohydrate-free formula with added maltodextrins
  Interventions: Other: Formula with maltodextrins
- Breastfeeding (No Intervention): Breastfed reference group

INTERVENTIONS:
Other: Formula with lactose
  Arms: Formula with lactose
Other: Formula with maltodextrins
  Arms: Formula with maltodextrins

SUMMARY:
The optimal choice of carbohydrate in infant formula needs to be assessed in more detail. Lactose has conventionally been used in most milk-based infant formulas, but more recently lactose-free formulas based on corn syrup solids/maltodextrins have gained in popularity. However, the metabolic consequences have not been examined.

In a pilot study, the investigators will assess the postprandial metabolic response to a meal of formula with either lactose or maltodextrins. A breastfed reference group is also included.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Term infants (gestational age 37-42 weeks)
* Birth weight 2500-4500g

Exclusion Criteria:

* Infant illness
* Maternal diabetes
* Maternal pregnancy complications

Ages: 3 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Glucose levels | 2 hours (Change from baseline to 15 min, 30 min, 60 min, 90 min and 120 min)
  The change in serum glucose levels are monitored following a test meal from baseline to 15 min, 30 min, 60 min, 90 min and 120 minutes

SECONDARY OUTCOMES:
Insulin levels | 2 hours (Change from baseline to 15 min, 30 min, 60 min, 90 min and 120 min)
  The change in plasma insulin levels are monitored following a test meal at baseline, 15 min, 30 min, 60 min, 90 min and 120 minutes
Metabolite levels | 2 hours (Change from baseline to 15 min, 30 min, 60 min, 90 min and 120 min)
  The change in plasma metabolite levels are monitored (using metabolomics) following a test meal at baseline, 15 min, 30 min, 60 min, 90 min and 120 minutes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Slupsky CM, He X, Hernell O, Andersson Y, Rudolph C, Lonnerdal B, West CE. Postprandial metabolic response of breast-fed infants and infants fed lactose-free vs regular infant formula: A randomized controlled trial. Sci Rep. 2017 Jun 16;7(1):3640. doi: 10.1038/s41598-017-03975-4. PMID 28623320